CLINICAL TRIAL: NCT05765448
Title: Effects of the Consumption of SEAweed Biomass Versus PROtein Isolates on Postprandial Satiety and Metabolism (The SEAPRO Study)
Brief Title: Effects of the Consumption of SEAweed Biomass Versus PROtein Isolates on Postprandial Satiety and Metabolism
Acronym: SEAPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022/00909
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Nutrition, Healthy
Keywords: alternative protein; postprandial satiety
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Non-blinded, randomised crossover trial with each participant testing 5 different test ingredients on 5 separate study sessions on 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Soy-based control meal (Active Comparator): Bowl of soup noodles prepared with 10g soy protein isolate soup base and consumed with a pack of plain crackers (approximately 65g available carbohydrate in total).
  Interventions: Other: Soy control
- Laver/nori macroalgae (Porphyra umbilicus) whole biomass-based treatment meal (Experimental): Bowl of soup noodles prepared with 10g Laver/nori macroalgae (Porphyra umbilicus) whole biomass soup base and consumed with a pack of plain crackers (approximately 65g available carbohydrate in total).
  Interventions: Other: Intervention (Laver/nori (Porphyra umbillicus) macroalgae whole biomass)
- Laver/nori macroalgae (Porphyra umbilicus) protein isolates-based treatment meal (Experimental): Bowl of soup noodles prepared with 10g Laver/nori macroalgae (Porphyra umbilicus) protein isolates soup base and consumed with a pack of plain crackers (approximately 65g available carbohydrate in total).
  Interventions: Other: Intervention (Laver/nori macroalgae (Porphyra umbillicus) protein isolates)
- Microalgae (Chlorella vulgaris) whole biomass-based treatment meal (Experimental): Bowl of soup noodles prepared with 10g microalgae (Chlorella vulgaris) whole biomass soup base and consumed with a pack of plain crackers (approximately 65g available carbohydrate in total).
  Interventions: Other: Intervention (Chlorella microalgae (Chlorella vulgaris) whole biomass)
- Microalgae (Chlorella vulgaris) protein isolates-based treatment meal (Experimental): Bowl of soup noodles prepared with 10g microalgae (Chlorella vulgaris) protein isolates soup base and consumed with a pack of plain crackers (approximately 65g available carbohydrate in total).
  Interventions: Other: Intervention (Chlorella microalgae (Chlorella vulgaris) protein isolates)

INTERVENTIONS:
Other: Soy control — Soy isolate control meal
  Arms: Soy-based control meal
Other: Intervention (Laver/nori (Porphyra umbillicus) macroalgae whole biomass) — Laver/nori (Porphyra umbillicus) macroalgae whole biomass treatment meal
  Arms: Laver/nori macroalgae (Porphyra umbilicus) whole biomass-based treatment meal
Other: Intervention (Laver/nori macroalgae (Porphyra umbillicus) protein isolates) — Laver/nori macroalgae (Porphyra umbillicus) protein isolates treatment meal
  Arms: Laver/nori macroalgae (Porphyra umbilicus) protein isolates-based treatment meal
Other: Intervention (Chlorella microalgae (Chlorella vulgaris) whole biomass) — Chlorella microalgae (Chlorella vulgaris) whole biomass treatment meal
  Arms: Microalgae (Chlorella vulgaris) whole biomass-based treatment meal
Other: Intervention (Chlorella microalgae (Chlorella vulgaris) protein isolates) — Chlorella microalgae (Chlorella vulgaris) protein isolates treatment meal
  Arms: Microalgae (Chlorella vulgaris) protein isolates-based treatment meal

SUMMARY:
There is a need to identify alternative sources of protein that can be introduced into diets to effectively meet the protein requirements of the population. Seaweed presents a potential source of sustainable, alternative protein. In order to determine their utility in future foods, in this study we will undertake an acute postprandial trial to explore whether a macroalgae (porphyra) and a microalgae (chlorella) protein isolates are more beneficial for acute metabolic health as compared to their respective whole biomasses. In particular, we will compare the effects of whole biomasses and their protein isolates on acute glucose homeostasis, amino acid availability as well as on satiety and gut hormones.

DETAILED DESCRIPTION:
Seaweed presents a potential source of sustainable, alternative protein. Broadly categorised into macroalgae and microalgae, macroalgae including those of the genus Porphyra are traditionally known as nori or laver and is a common ingredient in several Asian dishes such as soups and sushi. Porphyra is rich in protein, micronutrients and dietary fibre and the equivalent variety in New Zealand is a red macroalgae known as Karengo. A prominent genus of microalgae is Chlorella, which is a green microalgae also rich in protein and currently used mainly in dietary supplements. The interest in seaweed as an ingredient incorporated into meals, food products and dietary supplements has been growing due to their macronutrient composition and bioactive substances with studied health benefits including improvements in glucose homeostasis, appetite and anti-hypertensive and hypocholesterolemic properties.

However, controlled human studies comparing specific macroalgae and microalgae, particularly for their potential to be used as a source of alternative protein, has been limited. Therefore, the present study aims to compare macroalgae (Porphyra) biomass and its protein isolates versus microalgae (Chlorella) biomass and its protein isolates on postprandial satiety and nutrient metabolism in healthy adult Chinese males by adding these as ingredients to a noodle soup dish. We specifically aim to explore whether the protein isolates are superior to the respective whole biomasses in terms of glucose homeostasis, amino acid availability as well as in terms of satiety and gut hormones. Results from this study will be used towards future food applications to enhance the potential of the use of seaweed as a sustainable and nutritious source of alternative proteins.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese ethnicity
* Aged 21 to 50 years
* Able to give informed consent
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2

Exclusion Criteria:

* Diabetic (HbA1C ≥ 6.5%)
* Smoking
* Having a dislike towards seaweed- or soy-based products
* Having allergies or intolerances to any common food ingredients including seaweed, soy, eggs, seafood, fish, milk, peanuts, tree nuts, wheat, gluten, cereal, fruits, dairy products, meat, vegetables, sugar, sweeteners, natural food colourings or flavourings, etc.
* Following special diets or having intentional dietary restrictions (e.g, vegetarians/vegans)
* Not willing to adhere to diet modification as in the study protocol
* Taking part in strenuous physical activities
* Not willing to stop any strenuous activity during or within 24 hours of study days (for those actively participating in sports at the competitive and/or endurance levels)
* Having glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having alcohol consumption on > 4 days per week with ≥ 6 alcoholic drinks per week
* Having sustained elevation of blood pressure (≥140/90 mm Hg)
* Having previously undergone any gastrointestinal surgery or having history of gastrointestinal disorders
* Having a history of heart, liver, kidney, blood disorders (e.g., thalassemia) or thyroid dysfunctions
* Having history of tuberculosis, HIV, Hepatitis B or Hepatitis C infections
* Having any prescription medication or any other alternative medicines or supplements which may interfere with study measurements in the opinion of the study investigators
* Having donated blood within 4 weeks of study participation
* Having poor veins or having history of severe vasovagal syncope (blackouts or fainting) from blood draws

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Glucose | Up to 180 minutes
  Serum glucose measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes

SECONDARY OUTCOMES:
Insulin | Up to 180 minutes
  Serum insulin measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Triglycerides | Up to 180 minutes
  Serum triglycerides measured at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Amino acids | Up to 180 minutes
  Plasma amino acids measured at 0, 30, 60, 90, 120 and 180 minutes
GLP-1 | Time Frame: Up to 180 minutes
  Plasma GLP-1 measured at 0, 30, 60, 90, 120, 150 and 180 minutes
Ghrelin | Up to 180 minutes
  Plasma ghrelin measured at 0, 30, 60, 90, 120, 150 and 180 minutes
Satiety | Up to 180 minutes
  Satiety measured using VAS at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Hunger | Up to 180 minutes
  Hunger measured using VAS at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes
Gastrointestinal symptoms | Up to 180 minutes
  Gastrointestinal symptoms measured using gastrointestinal questionnaire at 0, 15, 60, 120 and 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No